CLINICAL TRIAL: NCT04929938
Title: Application of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders for Ultra High Risk for Psychosis Patients
Brief Title: Application of UP for Transdiagnostic Treatment of Emotional Disorders for UHR for Psychosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AR202003
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-12

CONDITIONS: Emotional Dysfunction; Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial in wich a group will receive inmediate UP plus standard intervention and the other one will be in a waiting list plus standard care at PIPPEP.
Who Masked: Outcomes Assessor
Masking Description: The evaluator will be blind to the condition that owns the patients included
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inmediate UP plus Treatment As Usual (Experimental): Treatment As Usual Plus Inmediate Virtual group Therapy applying the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders. The treatment consists in 15 weekly sessions of 120 minutes that combines cognitive-behavioural techniques to improve emotional self-regulation skills.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Waiting list plus Treatment As Usual (Active Comparator): A waiting list for treatment with delayed UP after 7 months while receiving the treatment as usual (WL + TAU).
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — This is a combination of cognitive-behavioural techniques oriented to improve the emotional regulation. The Unified Protocol is comprised of 8 modules and it is applied following The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders Manual (Barlow, 2017).

SUMMARY:
The principal aim of the study is to assess the efficacy of the Unified Protocol (UP) for the treatment of the comorbid symptomatology of patients with Ultra High Risk (UHR) for psychosis. The secondary aims would be to assess the effects of the intervention with the UP on the subthreshold positive symptoms and the transition to psychosis rates at 3 months follow-up, insight, positive and negative emotions, emotion regulation skills, personality, quality of life, cognitive distortions, psychosocial functioning and the maintenance of the effects at the 3 months of follow-up.

The study is a randomised controlled trial in which a group will receive inmediate UP plus standard intervention and the other one will be in a waiting list plus standard care at our Early Psychosis Program (PIPPEP).

The evaluator will be blind to the group that owns every patients. The sample will be 42 patients with UHR for psychosis with comorbid emotional symptoms and are visited at the PIPPEP of the CSMA Ripollet (PSSJD).

The assessment will be performed at baseline, at the end of treatment and at three months follow-up and will include: general psychopathology (SCID), anxiety and depression (BDI-II, BAI), positive and negative emotions (PANAS), emotional disregulation (DERS), personality (NEO-FFI), functionality (EEASL, MI), quality of life (QLI-sp), cognitive distortions (CBQ), insight (BCIS) and a scale of satisfaction created ad-hoc. At the end of each session with the UP we will assess depression and anxiety during the last week (ODSIS, OASIS). Treatment with the UP will consist in 15 group sessions of 8 patients, 120 minutes in addition to the treatment as usual.

DETAILED DESCRIPTION:
Main goal:

To evaluate the efficacy of UP in a group format for the treatment of comorbid symptoms present in UHR for psychosis.

Secondary goals:

1. Evaluate the effects of UP intervention on subthreshold positive symptoms
2. Evaluate the rates of transition to psychosis at 3 months in patients in the inmediate UP+TAU group intervention and compare them with those in the WL+TAU.
3. Evaluate the effect of UP treatment on quality of life.
4. Evaluate the effect of treatment on cognitive distortions and disease awareness.
5. Evaluate the effect of treatment on positive and negative emotions.
6. Evaluate the effect of treatment on emotion regulation skills.
7. Evaluate the effect of UP treatment on psychosocial functioning.
8. To know the levels of neuroticism and extraversion in UHR patients and to study if they constitute a modulating factor of the response to treatment with UP.
9. Evaluate in the medium term the maintenance of the effects of treatment with PU.
10. Evaluate the satisfaction of patients with the UP intervention.

The present study is a randomized controlled trial in which participants will be assigned to a treatment group that will receive immediate group treatment with UP in addition to the treatment as usual (UP + TAU) and the other group will be placed on a waiting list for treatment with delayed UP after 7 months while receiving the treatment as usual (WL + TAU).

The first group will receive immediate intervention with UP in online group format (UP + TAU) with a total of 15 sessions of 2 hours of weekly frequency in addition to the usual treatment in PIPPEP. The sessions will have a group format of 5-8 patients per group. An additional follow-up sessios will be held at 3 months after the end of the treatment sessions. The sessions will work on the 8 modules of UP for the transdiagnostic treatment of Emotional Disorders.

Treatment as usual on PIPPEP is a multidisciplinary treatment in which psychiatric sessions, nursing, social work and psychology are performed applying cognitive-behavioral psychotherapy. The frequency of visits can be weekly or fortnightly in the case of psychotherapy and the focus of the intervention would be the sub-threshold positive symptoms. Traditional cognitive-behavioral techniques such as behavioral experiments, cognitive restructuring, or exposure will be used as outlined in manuals created for this purpose. The usual duration of the visits will be one hour and the format will be individual.

Due to the restrictions arising from the pandemic situation by COVID-19, the group intervention will be in video conferencing format with a secure platform to maintain data protection. To ensure the adequacy of the GE intervention, the number of patients will be between 5-8.

The videoconferencing method will be secure and the personal data of the participants will be protected. The platform method that the Foundation San Joan de Deu will use is appropriate and contemplates the data protection regulations.

Patients will be randomized for inclusion in the experimental or control group using a list of random numbers and will be assigned according to the order of collection. The evaluator will be blind to the group to which the evaluated patient belongs.

Fidelity to the PU treatment protocol will be guaranteed through regular supervision with an accredited therapist.

The psychiatric medication prescribed for the patients in the study will be monitored, as well as any changes that may be made during the time of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of UHR for psychosis in the last 3 years and have been included in the Early Intervention of Psychosis Program.

3. Having comorbid emotional symptoms 4. Fluently speaking in spanish and/or catalan. 5. Sign informed consent (IC).

Exclusion Criteria:

1. Having a current or past frank psychotic episode.
2. Having an intellectual disability
3. Having an organic problem that better explains the symptoms presented by the subjects.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI-II) (Beck et al., 1996) | Baseline
  This self-applied scale consists of 21 items and assesses the severity (symptomatic intensity) of the depression with each item containing several self-assessment phrases.
Beck Depression Inventory (BDI-II) (Beck et al., 1996) | Immediatly after the intervention
  This self-applied scale consists of 21 items and assesses the severity (symptomatic intensity) of the depression with each item containing several self-assessment phrases.
Beck Depression Inventory (BDI-II) (Beck et al., 1996) | 3 month follow-up
  This self-applied scale consists of 21 items and assesses the severity (symptomatic intensity) of the depression with each item containing several self-assessment phrases.
Beck Anxiety Inventory (BAI) (Beck et al., 1993) | Baseline
  It is a self-applied scale of 21 items that assess the presence and severity of anxiety.
Beck Anxiety Inventory (BAI) (Beck et al., 1993) | Immediatly after the intervention
  It is a self-applied scale of 21 items that assess the presence and severity of anxiety.
Beck Anxiety Inventory (BAI) (Beck et al., 1993) | 3 months follow-up
  It is a self-applied scale of 21 items that assess the presence and severity of anxiety.
PANAS Positive and Negative Affectiveness Scale (Watson et al., 1988) | Baseline
  It is a self-administered scale consisting of 20 items that describe positive and negative emotions. Each item is answered with a 5-point Likert-type scale where 0 is the minimum score and 5 is the maximum.
PANAS Positive and Negative Affectiveness Scale (Watson et al., 1988) | Inmediatly after the intervention
  It is a self-administered scale consisting of 20 items that describe positive and negative emotions. Each item is answered with a 5-point Likert-type scale where 0 is the minimum score and 5 is the maximum.
PANAS Positive and Negative Affectiveness Scale (Watson et al., 1988) | 3 month follow-up
  It is a self-administered scale consisting of 20 items that describe positive and negative emotions. Each item is answered with a 5-point Likert-type scale where 0 is the minimum score and 5 is the maximum.
Scale of Severity and Deterioration of Depression (ODSIS) (Bentley et al., 2013) | Baseline
  This is a short 5-item questionnaire that continuously assesses the severity of symptoms and the deterioration of depression. Can be used in different depressive disorders
Scale of Severity and Deterioration of Depression (ODSIS) (Bentley et al., 2013) | Immediatly after the intervention
  This is a short 5-item questionnaire that continuously assesses the severity of symptoms and the deterioration of depression. Can be used in different depressive disorders
Scale of Severity and Deterioration of Depression (ODSIS) (Bentley et al., 2013) | 3 months follow-up
  This is a short 5-item questionnaire that continuously assesses the severity of symptoms and the deterioration of depression. Can be used in different depressive disorders
General Scale of Severity and Anxiety Impairment (OASIS) (Norman et al., 2006). | Baseline
  This is a short 5-item questionnaire that continuously assesses the severity of symptoms and deteriorating anxiety. Can be used in multiple anxiety disorders.
General Scale of Severity and Anxiety Impairment (OASIS) (Norman et al., 2006). | Immediatly after the intervention
  This is a short 5-item questionnaire that continuously assesses the severity of symptoms and deteriorating anxiety. Can be used in multiple anxiety disorders.
General Scale of Severity and Anxiety Impairment (OASIS) (Norman et al., 2006). | 3 months follow-up
  This is a short 5-item questionnaire that continuously assesses the severity of symptoms and deteriorating anxiety. Can be used in multiple anxiety disorders.
Difficulties in Emotion Regulation Scale (DERS) (Gratz et al., 2004) | Baseline
  It is a 28-item scale that measures emotional dysregulation in 5 dimensions:Non acceptance of Emotions, Difficulties Engaging in Goal-Directed Behavior When Distressed, Lack of Emotional Clarity, Lack of Emotional Awareness, Limited Access to Emotion Regulation Strategies and Impulse Control Difficulties.
Difficulties in Emotion Regulation Scale (DERS) (Gratz et al., 2004) | Inmediatly afther the intervention
  It is a 28-item scale that measures emotional dysregulation in 5 dimensions:Non acceptance of Emotions, Difficulties Engaging in Goal-Directed Behavior When Distressed, Lack of Emotional Clarity, Lack of Emotional Awareness, Limited Access to Emotion Regulation Strategies and Impulse Control Difficulties.
Difficulties in Emotion Regulation Scale (DERS) (Gratz et al., 2004) | 3 month follow-up
  It is a 28-item scale that measures emotional dysregulation in 5 dimensions:Non acceptance of Emotions, Difficulties Engaging in Goal-Directed Behavior When Distressed, Lack of Emotional Clarity, Lack of Emotional Awareness, Limited Access to Emotion Regulation Strategies and Impulse Control Difficulties.

SECONDARY OUTCOMES:
Socio-demographic questionnaire | Baseline
  This questionnaire collects basic information such as gender and clinical aspects like age of onset, number of admissions, treatment received and substance use.
Five Factor Personality Inventory (NEO-FFI) (Costa et al., 1999) | Baseline
  It is the reduced version of the NEO-PI-R and consists of 60 items that evaluate the personality according to 5 factors: Neuroticism, Extraversion, Openness, Kindness and Responsibility.
Five Factor Personality Inventory (NEO-FFI) (Costa et al., 1999) | 3 month follow-up
  It is the reduced version of the NEO-PI-R and consists of 60 items that evaluate the personality according to 5 factors: Neuroticism, Extraversion, Openness, Kindness and Responsibility.
Inadaptation Scale (EI) (Echeburúa et al., 2000). Resultados de traducción Scale of Inadaptation (EI) (Echeburúa et al. 2000) | Baseline
  It consists of 6 items that measure the impact that the current problems of the subjects have in different areas of their daily life (work, social life, leisure time, relationships, family life and globally).
Inadaptation Scale (EI) (Echeburúa et al., 2000). Resultados de traducción Scale of Inadaptation (EI) (Echeburúa et al. 2000) | Immediatly after the intervention
  It consists of 6 items that measure the impact that the current problems of the subjects have in different areas of their daily life (work, social life, leisure time, relationships, family life and globally).
Inadaptation Scale (EI) (Echeburúa et al., 2000). Resultados de traducción Scale of Inadaptation (EI) (Echeburúa et al. 2000) | 3 months follow-up
  It consists of 6 items that measure the impact that the current problems of the subjects have in different areas of their daily life (work, social life, leisure time, relationships, family life and globally).
Quality of Life Index (QLI-Sp) (Mezzich et al. 2000) | Baseline
  It is a 10-item questionnaire that assesses various aspects of health-related quality of life (physical disability, emotional well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, etc.). It is scored on a scale of 1-10 points, with the highest scores corresponding to a higher quality of life.
Quality of Life Index (QLI-Sp) (Mezzich et al. 2000) | Immediatly after the intervention
  It is a 10-item questionnaire that assesses various aspects of health-related quality of life (physical disability, emotional well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, etc.). It is scored on a scale of 1-10 points, with the highest scores corresponding to a higher quality of life.
Quality of Life Index (QLI-Sp) (Mezzich et al. 2000) | 3 months follow-up
  It is a 10-item questionnaire that assesses various aspects of health-related quality of life (physical disability, emotional well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, etc.). It is scored on a scale of 1-10 points, with the highest scores corresponding to a higher quality of life.
Cognitive Bias Questionnaire (CBQ) (Peters et al., 2013). | Baseline
  It consists of 30 statements which pose situations in the form of vignettes and measure the presence of 5 cognitive biases: intentionality, catastrophism, dichotomous thinking, hasty conclusions, and reasoning based on emotions.
Cognitive Bias Questionnaire (CBQ) (Peters et al., 2013). | Immediatly after the intervention
  It consists of 30 statements which pose situations in the form of vignettes and measure the presence of 5 cognitive biases: intentionality, catastrophism, dichotomous thinking, hasty conclusions, and reasoning based on emotions.
Cognitive Bias Questionnaire (CBQ) (Peters et al., 2013). | 3 months follow-up
  It consists of 30 statements which pose situations in the form of vignettes and measure the presence of 5 cognitive biases: intentionality, catastrophism, dichotomous thinking, hasty conclusions, and reasoning based on emotions.
Beck Cognitive Insight Scale (BCIS) (Beck et al., 2004) | Baseline
  It is a self-administered scale of 15 items with 4 response options. Collects information on the ability to correct erroneous judgments on two subscales: self-reflection and self-certainty.
Beck Cognitive Insight Scale (BCIS) (Beck et al., 2004) | Immediatly after the intervention
  It is a self-administered scale of 15 items with 4 response options. Collects information on the ability to correct erroneous judgments on two subscales: self-reflection and self-certainty.
Beck Cognitive Insight Scale (BCIS) (Beck et al., 2004) | 3 months follow-up
  It is a self-administered scale of 15 items with 4 response options. Collects information on the ability to correct erroneous judgments on two subscales: self-reflection and self-certainty.
The Treatment Opinion Scale (TSO) | Immediatly after the intervention
  This is a questionnaire created ad hoc to assess patients satisfaction with the treatment "Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders" created by Jorge Osma and collaborators in a Spanish sample of patients with Emotional Disorders of the public health system.
Mini International Neuropsychiatric Interview (MINI) 7.0.2. Spanish Version. (Sheehan, 2019) | Baseline
  This is a brief and high structured interview of the main psychiatric disorders of the IDC -10 and DSM-IV in order to be employed by psychiatrists and physicians not psychiatrists afterwards short time training.
Mini International Neuropsychiatric Interview (MINI) 7.0.2. Spanish Version. (Sheehan, 2019) | 3 months follow-up
  This is a brief and high structured interview of the main psychiatric disorders of the IDC -10 and DSM-IV in order to be employed by psychiatrists and physicians not psychiatrists afterwards short time training.
CAARMS (Yung et al., 2005). | Baseline
  It is a semi-structured interview that assesses subclinical psychotic symptoms in the previous year. The intensity and frequency of symptoms are recorded to distinguish between a non-risk state and a High Risk Mental State or a First Psychotic Episode.
CAARMS (Yung et al., 2005). | 3 months follow-up
  It is a semi-structured interview that assesses subclinical psychotic symptoms in the previous year. The intensity and frequency of symptoms are recorded to distinguish between a non-risk state and a High Risk Mental State or a First Psychotic Episode.

CONTACTS AND LOCATIONS:
Overall Officials: Trini Peláez, Principal Investigator — Parc Sanitari Sant Joan de Déu
Locations (2):
- Spain (2):
  - Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona
  - Fundació Sant Joan de Déu, Esplugues de Llobregat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelaez T, Lopez-Carrillero R, Ferrer-Quintero M, Ochoa S, Osma J. Application of the unified protocol for the transdiagnostic treatment of comorbid emotional disorders in patients with ultra-high risk of developing psychosis: A randomized trial study protocol. Front Psychol. 2022 Sep 1;13:976661. doi: 10.3389/fpsyg.2022.976661. eCollection 2022. PMID 36118431